Title of Research Study: Transcranial Direct Current Stimulation and Cognitive Remediation Therapy for Psychosis (IRB # 1311M45305)

## **Investigator Team Contact Information:**

For questions about research appointments, the research study, research results, or other concerns, call the study team at:

Investigator Name: Ian Ramsay, PhD Investigator Departmental Affiliation: Psychiatry & Behavioral Sciences Phone Number: 612-672-6805 Email Address: ramsa045@umn.edu

**Study Staff:** Areeb Kidwai Phone Number: 612-626-0953

Email Address: tdcsbraintrain@umn.edu

If your doctor is also the person responsible for this research study, please note that s/he is interested in both your clinical care and the conduct of this research study. You have the right to discuss this study with another person who is not part of the research team before deciding whether to participate in the research.

Supported By: This research is supported by the National Institute of Mental Health (NIMH) and the Frederick B. Wells, Jr. Schizophrenia Endowment Fund.

## **Key Information About This Research Study**

The following is a short summary to help you decide whether or not to be a part of this research study. More detailed information is listed later on in this form.

#### What is research?

Doctors and investigators are committed to your care and safety. There are important differences between research and treatment plans:

- The goal of research is to learn new things in order to help groups of people in the future. Investigators learn things by following the same plan with a number of participants, so they do not usually make changes to the plan for individual research participants. You, as an individual, may or may not be helped by volunteering for a research study.
- The goal of clinical care is to help you get better or to improve your quality of life. Doctors can make changes to your clinical care plan as needed.

 TEMPLATE LAST REVISED: 12/16/2019 Version Date:07Apr2022

## Why am I being asked to take part in this research study?

We are asking you to take part in this research study because you have been diagnosed with schizophrenia or schizoaffective disorder.

#### What should I know about a research study?

- Someone will explain this research study to you.
- Whether or not you take part is up to you.
- You can choose not to take part.
- You can agree to take part and later change your mind.
- Your decision will not be held against you.
- You can ask all the questions you want before you decide.

## Why is this research being done?

The purpose of this study is to evaluate the use of transcranial direct current stimulation (tDCS) and transcranial alternating current stimulation (tACS) for changing brain function. tDCS and tACS are experimental techniques used to stimulate the brain. The stimulation occurs outside the head. The procedure involves applying a small amount of electrical current across the scalp, for a short period of time. This small current is able to change the electrical activity inside the targeted areas of the brain. In our study, we will ask you to complete a series of computer based cognitive remediation sessions, while applying tDCS or tACS. We will also ask you to complete a series of cognitive tests to assess changes in brain speed, memory and attention. The information gained from this study will help us to understand how the brain works and how tDCS and tACS could be used to improve brain function.

tDCS and tACS (stimulation) involve applying a weak electrical current to the scalp. This study will use the Neuroelectrics Starstim device to apply stimulation. These devices are experimental and deliver the same type of stimulation. This device is experimental, meaning that it has not been approved by the FDA for use in this study. Instead, it is classified as a non-significant risk device for investigational (research) purposes.

## How long will the research last?

We expect that you will be in this research study for approximately two to three months.

#### What will I need to do to participate?

You will be asked to complete baseline assessments, participate in 10 brain training and stimulation sessions, complete post-training assessments, and complete follow-up assessments. Assessments include interviews about symptoms, questionnaires, cognitive tests, and EEGs.

More detailed information about the study procedures can be found under "What happens if I say yes, I want to be in this research?"

## Is there any way that being in this study could be bad for me?

The main risks of tDCS and tACS are minor and include headache, nausea, fatigue, dizziness, and itching, discomfort, and a burning sensation at the stimulation sites.

More detailed information about the risks of this study can be found under "What are the risks of this study? Is there any way being in this study could be bad for me? (Detailed Risks)" and in the "What


#### happens to the information collected for the research?" section

## Will being in this study help me in any way?

There are no benefits to you from your taking part in this research. We cannot promise any benefits to others from your taking part in this research. However, possible benefits to others include a better understanding of psychiatric conditions and the brain that could lead to improved therapies for psychiatric illnesses in the future.

## What happens if I do not want to be in this research?

You do not have to participate in this research. Instead of being in this research study, your choices may include:

- Participating in a commercially available cognitive training program
- Continuing your regular clinical care with your primary doctor/therapist

## **Detailed Information About This Research Study**

The following is more detailed information about this study in addition to the information listed above.

## How many people will be studied?

We expect about 105 people will be in this research study.

## What happens if I say "Yes, I want to be in this research"?

If you agree to participate in the study, we would ask you to do the following:

First, we would conduct a routine screening process to confirm that you are eligible to participate in this study. We would ask you questions about yourself, your mental health history, your symptoms, and how you are feeling.

If you are pregnant or become pregnant while on this study, please let the study team know right away. While there are no known risks associated with tDCS and tACS to pregnant women or fetuses, people who are pregnant or possibly pregnant will also be excluded from this study.

After the screening, you would be asked to continue participation in the study. Appointments are held at the University of Minnesota Medical Center (Fairview Riverside West Building) in the Department of Psychiatry's Ambulatory Research Center (ARC). During the COVID-19 pandemic, some research appointments may be held remotely using a video teleconferencing software called Zoom or through a phone call. At the first visit, study staff would interview you to gather demographic and health history information and ask you to complete a reading assessment and handedness questionnaire. The first visit with screening and other assessments would take approximately 2-2.5 hours. If you are enrolled in the Consortium of Psychosis Research Recruitment (COPRR), we may be able to use some data from previous studies to shorten the length of the first appointment. During 1-4 additional visits, you would be asked to complete several assessment using Electroencephalography (EEG) to measure brain waves would be completed. During the EEG you would be asked to participate in multiple tasks, which should take about 2-3 hours. These visits would take 6-9 hours in total.


Next, research staff would set up the stimulation device. The device consists of two saline soaked sponges beneath small electrodes. One sponge would be positioned on your scalp and the other sponge will be positioned on your forehead. You will then be asked to complete a series of computer-based tasks, which will last approximately 1 hour. The stimulation system will deliver a small electrical current through the saline soaked pads during the beginning of your computer-based task. The stimulation will then be turned off and you will complete the remainder of the computer-based task.

Half of the participants in this study will receive active stimulation during the training session. The other half of participants will receive sham stimulation, which will feel like active stimulation, but won't deliver meaningful electrical current during the whole training session. The treatment you get would be chosen by chance, like flipping a coin. Neither you nor the study doctor would choose what treatment you get. You would have a 50% chance of being given either treatment. Neither you nor the study staff will know which treatment you are getting.

If you become uncomfortable at any time during the session, or you experience a headache, please tell the experimenter and they will immediately stop the testing. A member of the research staff will constantly monitor each experiment to ensure your comfort and safety.

The total time involved in each experimental session would be between one and two hours. You would be asked to return 2-4 times per week for 3-5 weeks, for a total of 10 sessions. We would try to keep 24 hours between each stimulation session but can do multiple sessions in one day if necessary. After each session you would remain seated in the laboratory for at least 10 minutes after the stimulation has ended to be sure the risk of any short-term adverse effects, such as headache, have gone away.

After 5 training sessions, we would check in about some of your symptoms. This check-in would occur after a treatment session and would take approximately 5-10 minutes. Then after 10 sessions, you would complete assessments relating to cognition, feelings, symptoms, quality of life, social functioning, working memory, and the EEG assessments. These tasks would take approximately 5-8 hours over 1-4 appointments.

One month later, we would ask you to come back in for a follow-up appointment, where you would repeat those assessments (except for the EEG) one final time. There would be one additional brief assessment and you would be given a questionnaire that asks which treatment group you think you were placed in. In total, these assessments would take 2.5-3.5 hours and could be completed over 1-2 appointments.




In some cases, we may ask participants to come back to repeat visits. For example, the EEG device may not record all the data correctly. You do not have to repeat any visits if you do not want to.

Due to the quickly changing COVID-19 pandemic, we may need to abruptly stop conducting in-person appointments during your time in the study. If this happens, we will ask you to complete as many study procedures remotely (via Zoom or telephone call) as possible. If this happens and you are not able to complete certain in-person assessments (EEG, stimulation sessions), we will not be able to compensate


you for those assessments. There may be an opportunity to come back when in-person appointments resume to complete those assessments.

## What happens if I say "Yes", but I change my mind later?

If you take part in this research study, and want to leave, you should tell us. Your choice not to be in this study will not negatively affect your right to any present or future medical care, your academic standing as a student, or your present or future employment.

We will make sure that you stop the study safely. We will also talk to you about follow-up care, if needed.

If you stop being in the research, information about you that has already been collected may not be removed from the study database.

If you decide to leave the research, contact the study team so we know you would like to stop. We may ask you to participate in the end of treatment interview and the one month follow up interview, if you are willing to do so. However, you do not have to complete any more study activities once you decide to stop.

#### Can I be removed from the research?

It's possible that we will have to ask you to leave the study before you finish it. If this happens, we will tell you why. Possible reasons for removal include worsening mental health symptoms and adverse reactions to the study treatment. If we decide to stop the study treatment, we may still ask you to participate in the end of treatment and one month follow up appointments, although you do not have to participate in these activities if you don't want to.

# What are the risks of being in this study? Is there any way being in this study could be bad for me? (Detailed Risks)

tDCS/tACS Stimulation Risks: There are no significant risks associated with tDCS or tACS as reasonably anticipated. Adverse effects of tDCS and tACS are minor and may include headache, nausea, fatigue, itching, discomfort, burning sensation, dizziness, and a flashing sensation (phosphenes). Electrical currents used for stimulation in this study will be well within established safety limits and do not pose any harm to brain tissue. To further minimize this risk, we will exclude subjects with any personal history of seizures or epilepsy, metallic cranial plates, screws, or implanted device, history of craniotomy, eczema on the scalp, or pre-existing sores or lesions at the stimulation administration site. We will also exclude subjects with any known tumor or lesion in their brain, even without a history of seizures. There is also a very small risk of psychiatric changes following stimulation, which will be minimized by obtaining a positive and negative symptom scale and excluding subjects with an increase in symptoms during the experimental course. tDCS and tACS administration have been classified as non-significant risk procedures when administered by a trained professional and when proper safety screenings are in place. Like many procedures, the long-term effects are unknown. Overall, tDCS and tACS are considered safe procedures when administered by a trained professional and proper safety screenings are in place.


**Assessment risks:** You may experience some anxiety during the assessment tests in this study. It is good to keep in mind that there are many ways to answer any of the questions or tests, and there are no right or wrong answers. The questions and tests are used only to assess the effects of this study on how you feel, you're thinking, and your problem-solving skills.

You may feel tired or frustrated during the assessment testing or during the computerized training exercises. You are free to take breaks during some of the tests and activities. If you feel discomfort due to your participation, you may discontinue at any time.

**EEG Risks:** The gel applicator might feel rough and uncomfortable if you have sensitive skin on your scalp. The study staff will check in with you to make sure you aren't feeling too uncomfortable during the gel application. There is also a small risk of skin irritation from the electrode gel, although this is uncommon.

**Randomization risks:** You will be assigned to a treatment program (active tDCS or active tACS or sham stimulation) by chance, and the treatment you receive may prove to be less effective or to have more side effects than the other study treatment, or other available treatments.

Confidentiality: There is some risk of a data breach involving the information we have about you. We comply with the University's security standards to secure your information and minimize risks, but there is always a possibility of a data breach. Participation in research will involve a loss of privacy; however, your records will be handled as confidentially as possible. Dr. Ramsay, and his research staff will use a code when discussing your participation. They will not speak of you by name to anyone outside of the lab. Only Dr. Ramsay, his collaborators, and his assistants will have access to your tests and computerized training results. No identifying information will be used in any report or publications that may result from this study.

**Email Communications:** We will ask you to sign a separate consent form that contains information regarding email communication and its risks.

We will save emails that are sent to our email addresses as part of your study record. We will protect your emails as we do with any other records. We will remove your name, email address, and any other identifying information when we save your emails. However, you should think about the risks before sending emails with sensitive information (such as information about health conditions and symptoms).

**Texting:** We will ask you to sign a separate consent form that contains information regarding text communication and its risks.

We will not save text messages that are sent to us. They will be deleted with the conclusion of each conversation.

**COVID-19 Infection Risk:** Just like any in-person interaction, attending in-person research appointments comes with a risk of becoming infected with COVID-19. Some procedures will require close contact between you and our study staff. To lower the risk of spreading COVID-19, our staff will wear equipment designed to protect you and them from spreading germs. We will also require you to wear a mask while inside our buildings. In addition, staff will constantly be monitoring themselves for symptoms, all participants will be screened for symptoms and other risk factors before each appointment, participants


and staff will wash their hands before and after each appointment, social distancing will be enforced (when possible), and surfaces and equipment will be disinfected before and after each appointment. We imagine the risk of becoming infected with COVID-19 during study procedures is no more than the risk presented during an average trip to the grocery store. If you test positive for or experience symptoms of COVID-19 during the course of the study, please notify study staff immediately so proper precautions can be taken to reduce spread.

## Will it cost me anything to participate in this research study?

Taking part in this research study will not lead to any costs to you.

#### Will being in this study help me in any way? (Detailed Benefits)

There are no benefits to you from your taking part in this research. We cannot promise any benefits to others from your taking part in this research. However, possible benefits to others include a better understanding of psychiatric conditions and the brain that could lead to improved therapies for psychiatric illnesses in the future.

# What happens to the information collected for the research, including my health information?

We try to limit the use and sharing of your information, including research study records, any medical records and any other information about you, to people who have a need for this information. But we cannot promise complete confidentiality.

#### **Overview**

If you participate in this study, your information, including your health information, will be used and shared for purposes of conducting this research. As described later in this Consent Form, your information may also be used and shared for publishing and presenting the research results, future research, and any optional elements of the research you agree to in this Consent Form, which may include creating audio and video recordings of you. If you sign this Consent Form, you are giving us permission to use and share your health information for these purposes, and if we are using your medical records, you are giving permission to any health care providers who are treating you to share your medical records with us.

#### What health information will be made available?

Health information about you to be used and shared for the research includes those items checked by the research team below:

☐ Your medical records, which may include records from hospital and clinic visits, emergency room visits, immunizations, medical history and physical exams, medications, images and imaging reports, progress notes, psychological tests, EEG/EKG/ECHO reports, lab and pathology reports, dental records and/or financial records. These records may be used and shared for as long as this research continues.

☐ Information collected as part of this research study, including research procedures, research visits,


and any optional elements of the research you agree to, all as described in this Consent Form. This information might not be part of your medical record, and may include things like responses to surveys and questionnaires, and information collected during research visits described in this Consent Form.

#### What about more sensitive health information?

Some health information is so sensitive that it requires your specific permission. If this research study requires any of this sensitive information, the boxes below will be marked and you will be asked to initial to permit this information to be made available to the research team to use and share as described in this Consent Form.

| Who will access and use my health information? |
|--------------------------------------------------------------------|
| ☐ My sickle cell anemia records (initial) |
| ☑ My mental health diagnosis/treatment records (initial) |
| ☐ My genetic testing records (initial) |
| ☐ My HIV/AIDS testing records (initial) |
| ☐ My drug & alcohol abuse, diagnosis & treatment records (initial) |

If you agree to participate in this study, your information will be shared with:

- The University of Minnesota research team and any institutions or individuals collaborating on the research with us;
- Others at the University of Minnesota and M Health/Fairview who provide support for the
  research or who oversee research (such as the Institutional Review Board or IRB which is the
  committee that provides ethical and regulatory oversight of research at the University, systems
  administrators and other technical and/or administrative support personnel, compliance and
  audit professionals (Such as the Quality Assurance Program of the Human Research Protection
  Program (HRPP)), individuals involved in processing any compensation you may receive for your
  participation, and others);
- The research sponsor(s), any affiliates, partners or agents of the sponsor(s) involved in the research, organizations funding the research, and any affiliates, partners or agents of the funding organization(s) involved in the research;
  - National Institute of Mental Health (NIMH)
  - Frederick B. Wells, Jr. Schizophrenia Endowment Fund
- Organizations who provide accreditation and oversight for research and the research team, and
  others authorized by law to review the quality and safety of the research (such as U.S.
  government agencies like the Food and Drug Administration, the Office of Human Research
  Protections, the Office of Research Integrity, or government agencies in other countries); and


- Organizations that process any payments that may be made to you for participating in this study, and any other individuals or organizations specifically identified in this Consent Form.
  - Greenphire is the payment service we use to compensate you for your participation in this study. To register you in their system, we provide them with your full name, mailing address, and date of birth. All information collected and provided to Greenphire is stored in a secure fashion and will be kept confidential, except as required by law.
  - Posit Science Inc. has entered a Business Associate Agreement with the University of Minnesota to handle information for this research study and created the cognitive training software programs. Your data will be stored on their servers but will not have any identifying information.
  - VeraSci has entered a Data Use Agreement with the University of Minnesota to handle some assessment information for this research study. Your data will be stored on their servers but will not have any identifying information.

#### Additional sharing of your information for mandatory reporting

If we learn about any of the following, we may be required or permitted by law or policy to report this information to authorities:

- Current or ongoing child or vulnerable adult abuse or neglect;
- Communicable, infectious or other diseases required to be reported under Minnesota's Reportable Disease Rule;
- Certain wounds or conditions required to be reported under other state or federal law; or
- Excessive use of alcohol or use of controlled substances for non-medical reasons during pregnancy.

## How will my information be used in publications and presentations?

We may publish the results of this research in scientific, medical, academic or other journals or reports, or present the results at conferences. Information that makes it easy to identify you (such as your name and contact information, SSN and medical records number) will not be part of any publication or presentation. If you have an extremely unique or rare condition that is not shared by many others, it is possible that some people may be able to determine your identity even without these identifiers.

## What will be done with my data when this study is over?

We will use and may share data for future research. They may be shared with researchers/institutions outside of University of Minnesota. This could include for profit companies. We will not ask for your consent before using or sharing them. We will remove identifiers from your data and/or specimens, which means that nobody who works with them for future research will know who you are. Therefore, you will not receive any results or financial benefit from future research done on your specimens or data.

The sponsor, monitors, auditors, the IRB, the University of Minnesota Research Compliance Office and other University compliance units, the US Office of Research Integrity (ORI), the US Office for the


Protection of Human Research Protections (OHRP), the US Food and Drug Administration (FDA) may be granted direct access to your medical records to conduct and oversee the research. By signing this document you are authorizing this access. We may publish the results of this research. However, we will keep your name and other identifying information confidential.

A description of this clinical trial will be available at http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

# Do I have to sign this Consent Form and give my permission to make my information, including my health information, available for use and sharing?

No, you do not have to sign this Consent Form. But if you do not sign, you will not be able to participate in this research study. Treatment available outside of the study, payment for such treatment, enrollment in health insurance plans and eligibility for benefits will not be impacted by your decision about signing this Consent Form.

Does my permission for making my health information available for use and sharing ever expire?

No, there is no expiration date.

#### May I cancel my permission for making my health information available for use and sharing?

Yes. You may cancel your permission at any time by writing to the researcher at the address on the first page of this Consent Form. If you cancel your permission, you will no longer be in the research study. You may also want to ask someone on the research team in canceling will affect any research related medical treatment. If you cancel your permission, any health information about you that was already used and shared may continue to be used and shared for the research study and any optional elements of the study to which you agree in this Consent Form.

#### What happens to my health information after it is shared with others?

When we share your information with others as described in this Consent Form, privacy laws may no longer protect your information and there may be further sharing of your information.

#### Will I be able to look at my records?

It is possible that the research team may not allow you to see the information collected for this study. However, you may access any information placed in your medical records after the study is complete.

#### **Certificate of Confidentiality**

To help protect your privacy, the National Institutes of Health has granted a Certificate of Confidentiality. The researchers can use this Certificate legally to refuse to disclose information that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings, for example, if there is a court subpoena. The researchers will use the Certificate to resist any demands for information that would identify you, except as explained below.


The Certificate does not prevent a researcher from reporting information learned in research when required by other state or federal laws, such as mandatory reports to local health authorities for abuse or neglect of children/vulnerable adults, or information to the Food and Drug Administration (FDA) when required in an FDA audit. However, the Certificate limits the researcher from disclosing such information in follow up civil, criminal, legislative or administrative legal proceedings if the information was created or compiled for purposes of the research.

You also should understand that a Certificate of Confidentiality does not prevent you or a member of your family from voluntarily releasing information about yourself or your involvement in this research. If an insurer, medical care provider, or other person obtains your written consent to receive research information, then the researchers will not use the Certificate to withhold that information.

#### Will I receive research test results?

Most tests done on samples in research studies are only for research and have no clear meaning for health care. The investigator(s) will not contact you or share your individual test results.

## Will anyone besides the study team be at my consent meeting?

You may be asked by the study team for your permission for an auditor to observe your consent meeting. Observing the consent meeting is one way that the University of Minnesota makes sure that your rights as a research participant are protected. The auditor is there to observe the consent meeting, which will be carried out by the people on the study team. The auditor will not document any personal (e.g. name, date of birth) or confidential information about you. The auditor will not observe your consent meeting without your permission ahead of time.

## Whom do I contact if I have questions, concerns or feedback about my experience?

This research has been reviewed and approved by an IRB within the Human Research Protections Program (HRPP). To share feedback privately with the HRPP about your research experience, call the Research Participants' Advocate Line at 612-625-1650 (Toll Free: 1-888-224-8636) or go to z.umn.edu/participants. You are encouraged to contact the HRPP if:

- Your questions, concerns, or complaints are not being answered by the research team.
- You cannot reach the research team.
- You want to talk to someone besides the research team.
- You have questions about your rights as a research participant.
- You want to get information or provide input about this research.

#### Will I have a chance to provide feedback after the study is over?

The HRPP may ask you to complete a survey that asks about your experience as a research participant. You do not have to complete the survey if you do not want to. If you do choose to complete the survey, your responses will be anonymous.

If you are not asked to complete a survey, but you would like to share feedback, please contact the study team or the HRPP. See the "Investigator Contact Information" of this form for study team contact information and "Whom do I contact if I have questions, concerns or feedback about my experience?" of this form for HRPP contact information.


## What happens if I am injured while participating in this research?

In the event that this research activity results in an injury, treatment will be available, including first aid, emergency treatment and follow-up care as needed. Care for such injuries will be billed in the ordinary manner, to you or your insurance company. If you think that you have suffered a research related injury let the study investigators know right away.

## Will I be compensated for my participation?

If you agree to take part in this research study, we will pay you up to \$430 for your time and effort. The payment schedule is as follows:

Consent and diagnostic assessment: \$15

Baseline assessment completion: \$85

Treatment sessions: \$20 each \* 10 appointments = \$200

End of treatment assessment completion: \$85

One-month follow-up assessment: \$45

Payment will be made using a pre-paid debit card called Greenphire ClinCard. It works like a bank debit card. We will give you a debit card and each time you receive a payment for participation in this study, the money will be added to the card after each completed visit.

You may use this card at any store that accepts MasterCard or you can use a bank machine to remove cash. However, there may be fees drawn against the balance of the card for cash withdrawals (ATM use) and inactivity (no use for 6 months). We will give you the ClinCard Frequently Asked Questions information sheet that answers common questions about the debit card. You will also receive a cardholder agreement. Be sure to read all of this information for details about fees.

The debit card system is administered by an outside company. The company, Greenphire, and MasterCard, will be given your name and address. They will use this information only as part of the payment system. Your information will not be used for any other purposes and will not be given or sold to any other company. Greenphire and MasterCard will not receive any information about your health status or the study in which you are participating.

Additionally, you will have the option to receive updates related to appointment reminders and payment reminders and updates via text message and email message (Standard text messaging rates will apply). You will have the opportunity to opt-in to receive these messages, you are not required to provide your cell phone or email address to be enrolled in the study or use a ClinCard. If you choose to receive messages and decide at a later date that you want to stop these messages, you will have the ability to opt-out. If you choose to receive any communications via texts or emails, you will be asked to sign a separate form.

Payment you receive as compensation for participation in research is considered taxable income. If payment to an individual equals or exceeds \$600 in any one calendar year, the University of Minnesota is required to report this information to the Internal Revenue Service (IRS). Research payments to study participants that equal or exceed \$600 during any calendar year will result in a FORM 1099 (Miscellaneous Income) being issued to you and a copy sent to the IRS.


Discount tickets will be available to pay for your appointment parking expenses if you park in the ramps at the Fairview hospital location. At the end of each appointment, we can give you a discount ticket to cover the parking costs for the time you spent in the appointment with us. The researchers will not be able to compensate participants for any additional time spent parked in the ramps. You must be parked in a Fairview ramp for the researchers to cover your parking costs.

For other modes of transportation, you can receive up to \$100 in reimbursement throughout the study for public transportation or rides to appointments (taxi, Uber, Lyft, etc.). Receipts will be required for reimbursement of transportation costs and can be provided to the researchers in physical form (i.e. the paper receipt or a paper copy of it) or through email or text messaging.

## **Optional Elements:**

The following research activities are optional, meaning that you do not have to agree to them in order to participate in the research study. Please indicate your willingness to participate in these optional activities by placing your initials next to each activity.

| No,<br>I disagree | |
|---|---|
| | I give study staff permission to use data from and share data with the Consortium of Psychosis Research Recruitment (COPRR) if I am enrolled in it. |
| | I give the study staff permission to communicate about and set up my appointments using email. |
| | I give the study staff permission to communicate about and set up my appointments using text messaging. |
| | I give permission for study staff to contact my treating clinician to talk to them about the study and my clinical status. |
| | I would like to receive text and/or email alerts from Greenphire to alert me when funds are available on my ClinCard. |
| | The investigator may contact me in the future to see whether I am interested in participating in other research studies by Dr. Ian Ramsay. |
| ock for Capab<br>re documents<br>ocument. | le Adult: your permission to take part in this research. You will be provided a copy of |
| | I disagree |


| Signature of Participant | Date |
|------------------------------------------|------|
| Printed Name of Participant | |
| Signature of Person Obtaining Consent | Date |
| Printed Name of Person Obtaining Consent | |
